CLINICAL TRIAL: NCT03775512
Title: Evaluation of QDOT MICRO™ Catheter for Pulmonary Vein Isolation (PVI) in Subjects With PAF
Brief Title: Evaluation of QDOT MICRO™ Catheter for Pulmonary Vein Isolation in Subjects With Paroxysmal Atrial Fibrillation
Acronym: Q-FFICIENCY
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Biosense Webster, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Sequential | Masking: None | Purpose: Treatment
Other Study IDs: BWI_2017_07
Record Dates: First submitted 2018-11-23; First posted 2018-12-14 (Actual); Results first posted 2023-03-16 (Actual); Last update posted 2023-03-16 (Actual); Status verified 2023-02

CONDITIONS: Paroxysmal Atrial Fibrillation
MeSH Terms: conditions — Atrial Fibrillation

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: Yes | Unapproved Device: Yes

ARMS (2):
- Main Arm (Experimental): Subjects will be ablated with the QDOT Micro Catheter for Pulmonary Vein Isolation with nMARQ RF Generator
  Interventions: Device: RF Ablation with QDOT Micro
- Second Arm (variable flow) (Experimental): subjects will be treated with QDOT Micro catheter with variable flow nMARQ RF generator
  Interventions: Device: RF Ablation with QDOT Micro

INTERVENTIONS:
Device: RF Ablation with QDOT Micro — Subjects will be ablated using QDOT Micro catheter

SUMMARY:
Prospective, non-randomized, pre-market clinical evaluation of the QDOT MICRO™ Catheter to demonstrate the safety and effectiveness when compared to an historical control performance goal.

DETAILED DESCRIPTION:
Prospective, non-randomized, pre-market clinical evaluation of the QDOT MICRO™ Catheter to demonstrate the safety and effectiveness when compared to an historical control performance goal.

the trial has two arms: main arm and second arm (variable flow). The main arm will enroll 185 subjects and second arm will enroll 92 subjects.

ELIGIBILITY:
Key Inclusion Criteria:

* Symptomatic paroxysmal AF with one electrocardiographically documented AF episode within 6 months prior to enrollment and a a physician's note indicating recurrent self-terminating AF within 7 days . Documentation may include electrocardiogram (ECG); Transtelephonic monitoring (TTM), Holter monitor or telemetry strip.
* Failed at least one Class I or Class III antiarrhythmic drug as evidenced by recurrent symptomatic AF, contraindicated, or intolerable to the AAD.
* Age 18 years or older.

Key Exclusion Criteria:

* Previous surgical or catheter ablation for atrial fibrillation.
* AF secondary to electrolyte imbalance, thyroid disease, or reversible or non-cardiac cause.
* Previously diagnosed with persistent or long-standing persistent AF and/or Continuous AF > 7 days.
* Valve repair or replacement or presence of a prosthetic valve.
* CABG surgery within the past 6 months (180 days).
* Any carotid stenting or endarterectomy within the past 6 months.
* Coronary artery bypass grafting, cardiac surgery, or valvular cardiac surgical procedure within the past 6 months.
* Documented left atrium (LA) thrombus within 1 day prior to the index procedure.
* Documented LA size > 50 mm.
* Documented LVEF < 40%.
* Contraindication to anticoagulation (e.g., heparin).
* MI/PCI within the past 2 months.
* Documented thromboembolic event (including transient ischemic attack) within the past 12 months.
* Uncontrolled heart failure or New York Heart Association (NYHA) function class III or IV.
* Awaiting cardiac transplantation or other cardiac surgery within the next 12 months.
* Presence of implanted pacemaker or implantable cardioverter defibrillator (ICD).
* Women who are pregnant, lactating, or who are of child bearing age and plan on becoming pregnant during the course of the clinical investigation.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 283 (Actual)
Dates: Start 2019-01-30 (Actual); Primary Completion 2022-02-17 (Actual); Study Completion 2022-02-17 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Emile Daoud, Principal Investigator — Ohio State University; Jose Osorio, Principal Investigator — Grandview Medical Center; Francis Marchlinksi, Principal Investigator — University of Pennsylvania Health System; Michael Cutler, Principal Investigator — Intermountain Medical Center; Andrea Natale, Principal Investigator — Texas Cardiac Arrhythmia Research Foundation; Daniel Melby, Principal Investigator — Abbott Northwestern; Miguel Valderabanno, Principal Investigator — The Methodist Hospital Research Institute; George Monir, Principal Investigator — AdventHealth; Craig Delaughter, Principal Investigator — Texas Heart Health and Vascular; Christopher Liu, Principal Investigator — New York Presbyterian Hospital; Saumil Oza, Principal Investigator — Ascension St. Vincent's; Ayman Hussein, Principal Investigator — The Cleveland Clinic; Robert Fishel, Principal Investigator — JFK Hospital; Kenneth Ellenbogen, Principal Investigator — VCU; Gery Tomassoni, Principal Investigator — Baptist Hospital; Tristram Bahnson, Principal Investigator — Duke University; Chris Ellis, Principal Investigator — VUMC; Emerson Liu, Principal Investigator — Allegheny College; David Wilber, Principal Investigator — Loyola University; Moussa Mansour, Principal Investigator — Massachusetts General Hospital; Srinivas Dukkipati, Principal Investigator — Icahn School of Medicine at Mount Sinai; Hugh McElderry, Principal Investigator — University of Alabama at Birmingham; Ashish Patel, Principal Investigator — Wakemed Heart and Vascular; Larry Chinitz, Principal Investigator — NYU Langone Medical Center; Luigi DiBiase, Principal Investigator — Montefiore
Locations (22):
- United States (22):
  - Grandview Medical Center, Birmingham, Alabama
  - University of Alabama, Birmingham, Alabama
  - JFK Medical Center, Atlantis, Florida
  - Ascension St. Vincent's, Jacksonville, Florida
  - Florida Hospital, Orlando, Florida
  - Baptist Health, Lexington, Kentucky
  - Massachusetts General Hospital, Boston, Massachusetts
  - Abbott Northwestern Hospital Clinic, Minneapolis, Minnesota
  - NYU Langone, New York, New York
  - Mt. Sinai School of Medicine, New York, New York
  - New York Presbyterian Hospital, New York, New York
  - Montefiore Medical Center - Albert Einstein, The Bronx, New York
  - Duke University Medical Center, Durham, North Carolina
  - WakeMed Heart & Vascular, Raleigh, North Carolina
  - Cleveland Clinic, Cleveland, Ohio
  - Ohio State University, Columbus, Ohio
  - University of Penn Health System, Philadelphia, Pennsylvania
  - Texas Heart Health and Vascular, Arlington, Texas
  - St. David's - TCAR, Austin, Texas
  - Houston Methodist Hospital, Houston, Texas
  - Intermountain Medical Center, Murray, Utah
  - Virginia Commonwealth University, Richmond, Virginia

REFERENCES:
- [Derived] Osorio J, Hussein AA, Delaughter MC, Monir G, Natale A, Dukkipati S, Oza S, Daoud E, Di Biase L, Mansour M, Fishel R, Valderrabano M, Ellenbogen K; Q-FFICIENCY Trial Investigators. Very High-Power Short-Duration, Temperature-Controlled Radiofrequency Ablation in Paroxysmal Atrial Fibrillation: The Prospective Multicenter Q-FFICIENCY Trial. JACC Clin Electrophysiol. 2023 Apr;9(4):468-480. doi: 10.1016/j.jacep.2022.10.019. Epub 2023 Jan 18. PMID 36752484

RESULTS

PARTICIPANT FLOW:
Groups:
- Main Arm: QDOT Micro Catheter: Participants with symptomatic paroxysmal atrial fibrillation (PAF) who have failed at least one antiarrhythmic drug were ablated with electrophysiology mapping and radiofrequency (RF) ablation using QDOT Micro Catheter for pulmonary vein isolation with nMARQ radiofrequency (RF) generator.
- Variable Flow Arm: QDOT Micro Catheter: Participants with symptomatic PAF who have failed at least one antiarrhythmic drug were ablated with electrophysiology mapping and RF ablation using QDOT Micro Catheter for variable flow with nMARQ RF generator.
Period: Overall Study
Arm/Group | Main Arm: QDOT Micro Catheter | Variable Flow Arm: QDOT Micro Catheter
Started | 191 | 92
Treated | 177 | 87
Completed | 162 | 75
Not Completed | 29 | 17
Not completed — Death | 1 | 1
Not completed — Withdrawal by Subject | 7 | 4
Not completed — Lost to Follow-up | 5 | 5
Not completed — Excluded before Catheter insertion | 14 | 5
Not completed — Discontinued before RF energy applied on inserted catheter | 2 | 1
Not completed — Due to a late entrance criteria deviation | 0 | 1

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Main Arm: QDOT Micro Catheter | Variable Flow Arm: QDOT Micro Catheter | Total
Number analyzed (Participants) | 191 | 92 | 283
Age, Continuous [Mean (Standard Deviation); unit: years] | 63.5 (10.69) | 64.5 (9.75) | 64.0 (10.22)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 75 | 38 | 113
  Male | 116 | 54 | 170
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0
  Asian | 1 | 3 | 4
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 7 | 4 | 11
  White | 166 | 71 | 237
  More than one race | 0 | 0 | 0
  Unknown or Not Reported | 17 | 14 | 31

OUTCOME MEASURES:

1. Primary Outcome: Percentage of Participants With Early Onset Primary Adverse Events (PAEs): Atrio-esophageal Fistula and Pulmonary Vein (PV) Stenosis
Description: An adverse event (AE) is any untoward medical occurrence in a participant participating in a clinical study that does not necessarily have a causal relationship with the pharmaceutical/biological agent under study. A Primary AEs is an event which occurred within 90 days following initial and repeated ablation procedure using the QDOT MICRO. Primary AEs included: atrio-esophageal fistula and pulmonary vein stenosis.
Time Frame: Up to 90 days (post initial and repeated ablation procedure)
Population: The modified Intent-to-treat (mITT) analysis set included all enrolled participants who met all eligibility criteria and have the investigational device inserted.
Measure: Number; unit: Percentage of Participants
Arm/Group | Main Arm: QDOT Micro Catheter | Variable Flow Arm: QDOT Micro Catheter
Number analyzed (Participants) | 167 | 85
Percentage of Participants | 0 | 0

2. Primary Outcome: Percentage of Participants With Early Onset PAEs: Death, Myocardial Infraction, Cardiac Tamponade/Perforation, Thromboembolism, Stroke/Cardiovascular Accident , TIA, PNP, Heart Block, Pulmonary Edema, Vagal Nerve Injury, Pericarditis, and MVAC/Bleeding
Description: A Primary AEs is an event which occurred within the first week (7 days of the initial and repeated ablation procedure) which included death, myocardial infraction (MI), cardiac tamponade (CT)/perforation, thromboembolism, stroke/cardiovascular accident (CVA), transient ischemic attack (TIA), phrenic nerve paralysis (PNP), heart block, pulmonary edema, vagal nerve injury, pericarditis, and major vascular access complication/bleeding (MVAC).
Time Frame: Up to 7 days (post initial and repeated ablation procedure)
Population: The mITT analysis set included all enrolled participants who met all eligibility criteria and have the investigational device inserted.
Measure: Number; unit: Percentage of Participants
Arm/Group | Main Arm: QDOT Micro Catheter | Variable Flow Arm: QDOT Micro Catheter
Number analyzed (Participants) | 167 | 85
Percentage of Participants | 3.6 | 2.4

3. Primary Outcome: Percentage of Participants With Freedom From Documented Atrial Fibrillation (AF), Atrial Tachycardia (AT), or Atrial Flutter (AFL) Episodes or Other Failure Modes
Description: Percentage of participants with freedom from documented AF, AT, or AFL episodes or following failure modes: a) Acute procedural: Failure to confirm entrance block in all pulmonary veins post-procedure and use of a non-study catheter to treat left atrial ablation targets and Cavo-tricuspid isthmus; b) Repeat ablation: >2 repeat ablation procedures with the study catheter during the 3-Month blanking period (Day 0-90) after the index ablation procedure, use of a non-study catheter to treat study arrhythmia ablation targets during the blanking period, and any repeat ablation procedure during the Evaluation Period; c) Antiarrhythmic drug: taking a new AAD for AF or a previously failed AAD at a greater than the highest ineffective historical dose for AF during the evaluation period, were reported.
Time Frame: Day 91 to Day 365
Population: The per-protocol (PP) analysis set included participants who satisfied the following criteria: a) enrolled and meet eligibility criteria, b) had undergone RF ablation, c) were treated with the study catheters, and d) were treated for the study related arrhythmia, without major protocol deviations that deemed to affect the scientific integrity of the study. Here 'N' (number of participants analyzed) signifies the number of participants analyzed for this outcome measure.
Measure: Number; unit: Percentage of Participants
Arm/Group | Main Arm: QDOT Micro Catheter | Variable Flow Arm: QDOT Micro Catheter
Number analyzed (Participants) | 156 | 77
Percentage of Participants | 76.3 | 67.5

4. Secondary Outcome: Number of Participants With Unanticipated Adverse Device Effects (UADEs)
Description: Number of participants with UADEs were reported.
Time Frame: Up to 20 months
Population: The safety analysis set included all enrolled participants of the study who had the investigational device inserted, regardless if RF energy was delivered.
Measure: Count of Participants; unit: Participants
Arm/Group | Main Arm: QDOT Micro Catheter | Variable Flow Arm: QDOT Micro Catheter
Number analyzed (Participants) | 177 | 87
Participants | 0 | 0

5. Secondary Outcome: Number of Participants With Serious Non-Primary Adverse Events (SAEs) Within 7 Days (Early Onset), 8-30 Days (Peri-procedural) and Greater Than or Equal to (>=) 31 Days (Late Onset) of Initial Ablation Procedure
Description: Number of participants with serious non-primary AEs within 7 days (early onset), 8-30 days (peri-procedural) and >=31 days (late onset) of initial ablation were reported.
Time Frame: Within 7 days (early onset), 8-30 days (peri-procedural) and >=31 days (late onset) of initial ablation procedure (up to 20 months)
Population: as for outcome 4
Measure: Count of Participants; unit: Participants
Arm/Group | Main Arm: QDOT Micro Catheter | Variable Flow Arm: QDOT Micro Catheter
Number analyzed (Participants) | 177 | 87
Participants
  0 - 7 Days | 8 | 4
  8 - 30 Days | 4 | 3
  >= 31 Days | 25 | 12

6. Secondary Outcome: Number of Participants With Bleeding Complication by International Society on Thrombosis and Haemostasis (ISTH) Class and Timing of Onset
Description: Number of participants with bleeding complication (ISTH definitions): a) major, b) clinically relevant non-major and c) minor bleeding were reported. The ISTH classification of major bleeding event is a hemoglobin drop of greater than or equal to (>=) 2 grams per deciliter (g/dL), transfusion of >= 2 units (U) packed red blood cells, symptomatic bleed in a critical area, or fatal bleed. Clinically relevant non-major (CRNM) events require prolong hospitalization or result in laboratory testing, imaging, compression, procedure, interruption of the study medication or a change in concomitant therapy. Minor bleeding events are overt bleeding events that do not meet the criteria for CRNM or major bleeding events.
Time Frame: as for outcome 5
Population: as for outcome 4
Measure: Count of Participants; unit: Participants
Arm/Group | Main Arm: QDOT Micro Catheter | Variable Flow Arm: QDOT Micro Catheter
Number analyzed (Participants) | 177 | 87
Participants
  Major: 0 - 7 Days | 3 | 0
  Major: 8 - 30 Days | 0 | 0
  Major: >= 31 Days | 0 | 0
  CRNM: 0-7 Days | 3 | 0
  CRNM: 8-30 Days | 0 | 0
  CRNM: >= 31 Days | 2 | 0
  Minor: 0-7 Days | 5 | 0
  Minor: 8-30 Days | 1 | 0
  Minor: >= 31 Days | 2 | 0

7. Secondary Outcome: Percentage of Participants With Electrical Isolation of Pulmonary Veins (PVs) (Entrance Block) at the End of the Procedure
Description: Percentage of participants with electrical isolation of PVs (entrance block) at the end of the procedure were reported
Time Frame: End of the Procedure (up to 20 months)
Population: The PP analysis set included participants who satisfied the following criteria: a) enrolled and meet eligibility criteria, b) had undergone RF ablation, c) were treated with the study catheters, and d) were treated for the study related arrhythmia, without major protocol deviations that deemed to affect the scientific integrity of the study. Here 'N' (number of participants analyzed) signifies the number of participants analyzed for this outcome measure.
Measure: Number; unit: Percentage of Participants
Arm/Group | Main Arm: QDOT Micro Catheter | Variable Flow Arm: QDOT Micro Catheter
Number analyzed (Participants) | 164 | 82
Percentage of Participants | 100 | 100

8. Secondary Outcome: Percentage of Participants With Electrical Isolation of PV After First Encirclement With Acute Reconnection
Description: Percentage of participants with electrical isolation of PV after first encirclement with acute reconnection were reported.
Time Frame: Up to 20 months
Population: as for outcome 7
Measure: Number; unit: Percentage of Participants
Arm/Group | Main Arm: QDOT Micro Catheter | Variable Flow Arm: QDOT Micro Catheter
Number analyzed (Participants) | 164 | 82
Percentage of Participants | 42.7 | 31.7

9. Secondary Outcome: Percentage of Participants With Electrical Isolation of PV After First Encirclement Without Acute Reconnection
Description: Percentage of participants with electrical isolation of PV after first encirclement without acute reconnection were reported.
Time Frame: Up to 20 months
Population: as for outcome 7
Measure: Number; unit: Percentage of Participants
Arm/Group | Main Arm: QDOT Micro Catheter | Variable Flow Arm: QDOT Micro Catheter
Number analyzed (Participants) | 164 | 82
Percentage of Participants | 57.3 | 68.3

10. Secondary Outcome: Percentage of Participants With Pulmonary Veins (PV) Touch-up
Description: Percentage of participants with PV touch-up were reported. PV touch-up was defined as additional ablations being performed after first encirclement for targeted veins with acute reconnection.
Time Frame: Up to 20 months
Population: as for outcome 7
Measure: Number; unit: Percentage of Participants
Arm/Group | Main Arm: QDOT Micro Catheter | Variable Flow Arm: QDOT Micro Catheter
Number analyzed (Participants) | 164 | 82
Percentage of Participants | 42.7 | 31.7

11. Secondary Outcome: Percentage of Targeted Veins With Touch-up (Ablation of Acute Reconnection) Among All Targeted Veins
Description: Percentage of targeted veins with touch-up (ablation of acute reconnection) among all targeted veins were reported.
Time Frame: Up to 20 months
Population: as for outcome 7
Measure: Number; unit: Percentage of Targeted Veins
Units Other Than Participants: Targeted Veins
Arm/Group | Main Arm: QDOT Micro Catheter | Variable Flow Arm: QDOT Micro Catheter
Number analyzed (Participants) | 164 | 82
Number analyzed (Targeted Veins) | 328 | 164
Percentage of Targeted Veins | 27.4 | 20.7

12. Secondary Outcome: Percentage of Participants With Touch-up at Anatomical Location of Acute PV Reconnection After First Encirclement
Description: Percentage of participants with touch-up at anatomical location of acute PV reconnection after first encirclement was reported. The location included anterior, superior, ridge, posterior, and inferior region of the left pulmonary veins (LPV) and right pulmonary veins (RPV). The review of all ablation targets for the 1 participant with RPV ridge entered by site resulted in reclassification to RPV superior. This outcome measure was planned to be analyzed for specified arm (main arm) only.
Time Frame: Up to 20 months
Population: The PP set had participants who satisfied these criteria: a) enrolled and meet eligibility criteria, b) had undergone RF ablation, c) treated with the study catheters, and d) were treated for the study related arrhythmia, without major protocol deviations that deemed to affect the scientific integrity of the study. Here 'N' (number of participants analyzed) is number of participants analyzed for this endpoint and 'n' (number analyzed) is number of participants analyzed for specified categories.
Measure: Number; unit: Percentage of Participants
Arm/Group | Main Arm: QDOT Micro Catheter
Number analyzed (Participants) | 45
Percentage of Participants
  LPV: Anterior | 31.1
  LPV: Inferior | 28.9
  LPV: Posterior | 53.3
  LPV: Ridge | 42.2
  LPV: Superior | 44.4
  RPV: Anterior: number analyzed (Participants) | 43
  RPV: Anterior | 53.5
  RPV: Inferior: number analyzed (Participants) | 43
  RPV: Inferior | 37.2
  RPV: Posterior: number analyzed (Participants) | 43
  RPV: Posterior | 58.1
  RPV: Superior: number analyzed (Participants) | 43
  RPV: Superior | 27.9

13. Secondary Outcome: Percentage of Participants Who Underwent Repeat Ablation Procedures
Description: Percentage of participants who underwent repeat ablation procedures were reported.
Time Frame: Up to 20 months
Population: The PP analysis set included participants who satisfied the following criteria: a) enrolled and meet eligibility criteria, b) had undergone RF ablation, c) were treated with the study catheters, and d) were treated for the study related arrhythmia, without major protocol deviations that deemed to affect the scientific integrity of the study.
Measure: Number; unit: Percentage of Participants
Arm/Group | Main Arm: QDOT Micro Catheter | Variable Flow Arm: QDOT Micro Catheter
Number analyzed (Participants) | 166 | 82
Percentage of Participants | 10.8 | 13.4

14. Secondary Outcome: Percentage of Participants With PVs Re-isolation Among All of the Targeted PVs at Repeat Procedure
Description: Percentage of participants with PVs re-isolation among all of the targeted PVs at repeat procedure were reported.
Time Frame: Up to 20 months
Population: as for outcome 7
Measure: Number; unit: Percentage of Participants
Arm/Group | Main Arm: QDOT Micro Catheter | Variable Flow Arm: QDOT Micro Catheter
Number analyzed (Participants) | 23 | 11
Percentage of Participants | 100 | 100

15. Secondary Outcome: Percentage of Participants Requiring New Linear Lesion and/or New Foci Identified During the Repeat Ablation Procedure
Description: Percentage of participants requiring new linear lesion and/or new foci identified during the repeat ablation procedure were reported.
Time Frame: Up to 20 months
Population: as for outcome 7
Measure: Number; unit: Percentage of Participants
Arm/Group | Main Arm: QDOT Micro Catheter | Variable Flow Arm: QDOT Micro Catheter
Number analyzed (Participants) | 18 | 11
Percentage of Participants | 50.0 | 63.6

16. Secondary Outcome: Percentage of Participants With 12-Month Single Procedure Success
Description: Percentage of participants with 12-month single procedure success were reported. The 12-month single procedure success is defined as freedom from documented AF/AFL/AT recurrence (episodes > 30 seconds) during the evaluation period after a single ablation procedure.
Time Frame: Up to 12 months
Population: as for outcome 13
Measure: Number; unit: Percentage of Participants
Arm/Group | Main Arm: QDOT Micro Catheter | Variable Flow Arm: QDOT Micro Catheter
Number analyzed (Participants) | 166 | 82
Percentage of Participants | 77.3 | 72.4

ADVERSE EVENTS:
Time Frame: Up to 20 months
Description: The safety analysis set included all enrolled participants who had the investigational device inserted, regardless if RF energy was delivered.
Arm/Group | Main Arm: QDOT Micro Catheter | Variable Flow Arm: QDOT Micro Catheter
All-Cause Mortality (participants affected / at risk) | 1/177 | 1/87
Serious Adverse Events (participants affected / at risk) | 32/177 | 14/87
Other Adverse Events (participants affected / at risk) | 58/177 | 19/87
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Main Arm: QDOT Micro Catheter (N=177) | Variable Flow Arm: QDOT Micro Catheter (N=87)
Atrial fibrillation (Cardiac disorders) | 14 (16) | 6 (6)
Atrial flutter (Cardiac disorders) | 8 (8) | 4 (4)
Cardiac failure congestive (Cardiac disorders) | 2 (2) | 2 (2)
Cardiac tamponade (Cardiac disorders) | 2 (2) | 0 (0)
Chest pain (General disorders) | 6 (6) | 0 (0)
Pyrexia (General disorders) | 2 (2) | 0 (0)
Arteriovenous fistula (Vascular disorders) | 2 (2) | 0 (0)
Pleuritic pain (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 2 (2)
Sinus node dysfunction (Cardiac disorders) | 0 (0) | 2 (2)
Cardiac valve fibroelastoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 2 (2)
Headache (Nervous system disorders) | 1 (1) | 4 (4)
Migraine (Nervous system disorders) | 0 (0) | 3 (3)
Pericardial effusion (Cardiac disorders) | 2 (2) | 0 (0)
Pulmonary embolism (Respiratory, thoracic and mediastinal disorders) | 2 (2) | 0 (0)
Cardiac failure (Cardiac disorders) | 0 (0) | 2 (2)
Thrombocytopenia (Blood and lymphatic system disorders) | 2 (2) | 0 (0)
Angina unstable (Cardiac disorders) | 2 (2) | 2 (2)
Atrial tachycardia (Cardiac disorders) | 2 (2) | 4 (4)
Atrioventricular block (Cardiac disorders) | 2 (2) | 0 (0)
Cardiac arrest (Cardiac disorders) | 2 (2) | 0 (0)
Tachycardia (Cardiac disorders) | 4 (4) | 0 (0)
Ventricular extrasystoles (Cardiac disorders) | 2 (2) | 0 (0)
Cyst (General disorders) | 2 (2) | 0 (0)
Prostate cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 2 (2) | 0 (0)
Syncope (Nervous system disorders) | 1 (1) | 0 (0)
Transient ischemic attack (Nervous system disorders) | 1 (1) | 0 (0)
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 2 (2) | 0 (0)
Aortic dilatation (Vascular disorders) | 2 (2) | 0 (0)
Orthostatic hypotension (Vascular disorders) | 2 (2) | 0 (0)
Abdominal pain (Gastrointestinal disorders) | 2 (2) | 0 (0)
Gastrointestinal hemorrhage (Gastrointestinal disorders) | 2 (2) | 0 (0)
Hiatus hernia (Gastrointestinal disorders) | 2 (2) | 0 (0)
Abscess (Infections and infestations) | 2 (2) | 0 (0)
Diverticulitis (Infections and infestations) | 2 (2) | 0 (0)
Pneumonia (Infections and infestations) | 4 (4) | 0 (0)
Vascular pseudoaneurysm (Injury, poisoning and procedural complications) | 2 (2) | 0 (0)
Arthropathy (Musculoskeletal and connective tissue disorders) | 2 (2) | 0 (0)
Bursitis (Musculoskeletal and connective tissue disorders) | 2 (2) | 0 (0)
Nephrolithiasis (Renal and urinary disorders) | 2 (2) | 0 (0)
Aortic valve calcification (Cardiac disorders) | 0 (0) | 2 (2)
Cardiovascular disorder (Cardiac disorders) | 0 (0) | 2 (2)
Retroperitoneal haemorrhage (Gastrointestinal disorders) | 0 (0) | 2 (2)
Chest discomfort (General disorders) | 0 (0) | 2 (2)
Corona virus infection (Infections and infestations) | 0 (0) | 2 (2)
Hip fracture (Injury, poisoning and procedural complications) | 0 (0) | 2 (2)
Haemorrhagic stroke (Nervous system disorders) | 0 (0) | 2 (2)
Peripheral vascular disorder (Vascular disorders) | 0 (0) | 2 (2)
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Main Arm: QDOT Micro Catheter (N=177) | Variable Flow Arm: QDOT Micro Catheter (N=87)
Cardiac Tamponade/Perforation (Cardiac disorders) | 2 (2) | 1 (1)
Phrenic Nerve Injury / Diaphragmatic Paralysis (Nervous system disorders) | 1 (2) | 0 (0)
Major Vascular Access Complication / Bleeding (Vascular disorders) | 3 (3) | 0 (0)
Pulmonary Edema (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1)
Pericardial effusion (Cardiac disorders) | 4 (4) | 2 (2)
Angina pectoris (Cardiac disorders) | 2 (2) | 0 (0)
Atrial flutter (Cardiac disorders) | 4 (4) | 0 (0)
Pericarditis (Cardiac disorders) | 4 (4) | 0 (0)
Vomiting (Gastrointestinal disorders) | 2 (2) | 0 (0)
Chest pain (General disorders) | 2 (2) | 0 (0)
Non-Cardiac Chest pain (General disorders) | 4 (4) | 0 (0)
Urinary tract infection (Infections and infestations) | 2 (2) | 0 (0)
Incision site hemorrhage (Injury, poisoning and procedural complications) | 2 (2) | 0 (0)
Urinary tract injury (Injury, poisoning and procedural complications) | 2 (2) | 0 (0)
Laboratory test abnormal (Investigations) | 2 (2) | 0 (0)
Weight increased (Investigations) | 2 (2) | 0 (0)
Groin pain (Musculoskeletal and connective tissue disorders) | 2 (2) | 0 (0)
Joint swelling (Musculoskeletal and connective tissue disorders) | 2 (2) | 0 (0)
Musculoskeletal chest pain (Musculoskeletal and connective tissue disorders) | 2 (2) | 0 (0)
Neck Pain (Musculoskeletal and connective tissue disorders) | 2 (2) | 0 (0)
Headache (Nervous system disorders) | 5 (5) | 0 (0)
Hypoesthesia (Nervous system disorders) | 2 (2) | 0 (0)
Migraine (Nervous system disorders) | 2 (2) | 0 (0)
Presyncope (Nervous system disorders) | 2 (2) | 0 (0)
Hematuria (Renal and urinary disorders) | 3 (3) | 2 (2)
Prostatitis (Reproductive system and breast disorders) | 2 (2) | 0 (0)
Dyspnea (Respiratory, thoracic and mediastinal disorders) | 8 (8) | 0 (0)
Oropharyngeal pain (Respiratory, thoracic and mediastinal disorders) | 3 (3) | 0 (0)
Pleuritic pain (Respiratory, thoracic and mediastinal disorders) | 2 (2) | 0 (0)
Hematoma (Vascular disorders) | 2 (2) | 4 (4)
Hypertension (Vascular disorders) | 2 (2) | 8 (10)
Hypotension (Vascular disorders) | 12 (12) | 0 (0)
Fluid overload (Metabolism and nutrition disorders) | 2 (2) | 2 (2)
Vaginal hemorrhage (Reproductive system and breast disorders) | 2 (2) | 0 (0)
Pulmonary vein stenosis (Respiratory, thoracic and mediastinal disorders) | 6 (6) | 0 (0)
Atrial tachycardia (Cardiac disorders) | 4 (4) | 2 (2)
Coronary artery disease (Cardiac disorders) | 1 (1) | 2 (2)
Palpitations (Cardiac disorders) | 1 (1) | 0 (0)
Sinus bradycardia (Cardiac disorders) | 2 (2) | 0 (0)
Sinus tachycardia (Cardiac disorders) | 2 (2) | 0 (0)
Supraventricular extrasystoles (Cardiac disorders) | 4 (4) | 2 (2)
Supraventricular tachycardia (Cardiac disorders) | 6 (6) | 4 (4)
Ventricular arrhythmia (Cardiac disorders) | 2 (2) | 0 (0)
Ventricular extrasystoles (Cardiac disorders) | 8 (8) | 2 (2)
Ventricular tachycardia (Cardiac disorders) | 4 (4) | 0 (0)
Peripheral swelling (General disorders) | 2 (2) | 0 (0)
Heart rate increased (Investigations) | 2 (2) | 0 (0)
Carotid artery stenosis (Nervous system disorders) | 2 (2) | 0 (0)
Seizure (Nervous system disorders) | 2 (2) | 0 (0)
Pleural effusion (Respiratory, thoracic and mediastinal disorders) | 2 (2) | 0 (0)
Epistaxis (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0)
Fatigue (General disorders) | 0 (0) | 2 (2)
Anaesthetic complication (Injury, poisoning and procedural complications) | 0 (0) | 2 (2)
Procedural haemorrhage (Injury, poisoning and procedural complications) | 0 (0) | 2 (2)
Orthostatic hypotension (Vascular disorders) | 0 (0) | 2 (2)
Dizziness (Nervous system disorders) | 0 (0) | 2 (2)
Tachycardia (Cardiac disorders) | 0 (0) | 2 (2)
Abdominal distension (Gastrointestinal disorders) | 0 (0) | 2 (2)
Hypokalaemia (Metabolism and nutrition disorders) | 0 (0) | 2 (2)
Chronic obstructive pulmonary disease (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 4 (4)
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 2 (2)
Dyspnoea exertional (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 2 (2)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
Publications and presentation of clinical investigation results will be coordinated between sponsor and the clinical investigation authors. Authorship to be determined prior to development of any manuscript. All information concerning the study, investigational medical device, sponsor operations, patent application, manufacturing processes and basic scientific data supplied by the sponsor to the investigator and not previously published, are confidential and remain sole property of the sponsor.

DOCUMENTS (2):
  • Study Protocol (2021-02-03): https://cdn.clinicaltrials.gov/large-docs/12/NCT03775512/Prot_000.pdf
  • Statistical Analysis Plan (2021-07-22): https://cdn.clinicaltrials.gov/large-docs/12/NCT03775512/SAP_001.pdf